CLINICAL TRIAL: NCT00934297
Title: Evaluation of a New Multi-modality Visualization Tool for Investigation of Breast Lesions
Brief Title: Visualization Tool for Investigation of Breast Lesions
Status: Terminated | Type: Observational
Why Stopped: The study was terminated as the PI left the institution.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. Petrina Causer, Sunnybrook Health Sciences Centre
Other Study IDs: 049-2009
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Breast Lesions
Keywords: MRI visible breast lesions that are occult under ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pilot group: Real-time US imaging with simultaneous display of dynamically corresponding MR images (from a previous MRI screening) will be used to re-locate the lesion previously reported as occult under a second-look ultrasound screening.

SUMMARY:
Magnetic resonance imaging (MRI) is commonly used for the detection of breast lesions in genetically high-risk women due to its high sensitivity. As non-cancerous conditions including normal changes due to a woman's menstrual cycle may have the appearance of cancer on MR images, a biopsy (generally performed under ultrasound-guidance) of the suspicious mass is required for definitive diagnosis. However, only a limited percentage of MRI-visible lesions are also visible on ultrasound (US). Even if found, it is often unclear whether the lesion identified on US corresponds to the MRI-detected lesion in question. The investigators have developed a visualization tool to assist the visualization of MRI-detected lesions in US-guided procedures (e.g., biopsy). This tool provides a simultaneous display of the previously acquired MRI data alongside real-time US images. The investigators propose a pilot study to assess the usefulness of this tool in identifying MRI-detected lesions using real-time US-guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MRI-identified lesions that cannot be visualized under the second-look ultrasound examination, and who will undergo the recommended unilateral MRI follow-up.

Exclusion Criteria:

* US-visible lesion.
* Any contraindications to MRI (e.g., pacemakers, metal implants).
* Any contraindications to US imaging.
* Pregnancy.
* Claustrophobia.
* Inability to lie still for 45 minutes-1 hour.
* In excess of 250 pounds.
* Incapability to provide informed consent.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients clinically suspicious for breast cancer will undergo the standard bilateral MRI protocol, with the patient in the prone position and both breasts immobilized. Patients with a BIRADS reading of 4 or 5 based on the initial MRI are called back for a second-look US examination to determine if the lesion can be found using US imaging. If the lesion is occult to US during this second-look examination, the radiologist may recommend a follow-up high-resolution unilateral MRI to further characterize the lesion.
  For this feasibility study, 10 patients with MRI-identified lesions that cannot be visualized under the second-look ultrasound examination, and who will undergo the recommended unilateral MRI follow-up will be asked to participate in our research study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Target identification success: this outcome measure is a 'yes/no' outcome, indicating whether or not an MRI-detected lesion could be successfully visualized using US-guidance in the supplemental US exam | Time of examination

SECONDARY OUTCOMES:
Confidence scale for lesion visualization This is a 5-point scale: 1 - very low confidence; 2 - low confidence; 3 - ambiguous; 4 - confident; 5 - very confident | Time of examination

CONTACTS AND LOCATIONS:
Overall Officials: Petrina Causer, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada